CLINICAL TRIAL: NCT02308566
Title: Aortic Valve Replacement Using Closed Extracorporeal Circuit. Minimized Versus Conventional Extracorporeal Circulation Technique: Qualitative Differences
Brief Title: Cerebral Embolic Load in Patients Undergoing Surgical Aortic Valve Replacement: A Comparison of the Conventional With the Minimized Extracorporeal Circulation Technique Using Transcranial Doppler Ultrasound
Acronym: AKE-MECC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 034/11
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Aortic Valve Stenosis; Extracorporeal Circulation
Keywords: Intracranial Embolism; Ultrasonography, Doppler, Transcranial
MeSH Terms: conditions — Aortic Valve Stenosis; Intracranial Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Extracorporeal Circulation Technique (Active Comparator): Conventional Extracorporeal Circulation Technique
  Interventions: Procedure: Conventional Extracorporeal Circulation (CECC)
- Minimized Extracorporeal Circulation Technique (Experimental): Minimized Extracorporeal Circulation Technique
  Interventions: Procedure: Minimized Extracorporeal Circulation (MECC)

INTERVENTIONS:
Procedure: Minimized Extracorporeal Circulation (MECC) — This group of patients receives surgical aortic valve replacement using MECC.
  Arms: Minimized Extracorporeal Circulation Technique
Procedure: Conventional Extracorporeal Circulation (CECC) — This group of patients receives surgical aortic valve replacement using CECC.
  Arms: Conventional Extracorporeal Circulation Technique

SUMMARY:
In this study, the investigators aim to compare cerebral embolic load in patients undergoing surgical aortic valve replacement using either the minimized extracorporeal circulation or the conventional extracorporeal circulation technique. The detection of cerebral emboli is performed not-invasively by transcranial Doppler detection of high-intensity transient signals representing solid or gaseous microembolism in the middle cerebral arteries. The investigators hope to get more insight in the mechanism (incl. quantity) of cerebral embolism during aortic valve surgery using extracorporeal circulation.

DETAILED DESCRIPTION:
Background

The gold standard to treat severe aortic valve stenosis is currently the surgical aortic valve replacement (SAVR) using conventional extracorporeal circulation (CECC). SAVR, however, can be performed also on minimized extracorporeal circulation (MECC), which is characterized by reduced priming volume and interfaces between blood and artificial surfaces and blood-air interface, respectively. Further technical developments of the MECC system together with reports on less induction of the coagulation cascade and activation of inflammatory systemic response may account for a reduced incidence of microbubble generation with MECC system.

Objective

The aim of the is to investigate the procedural-related incidence of high-intensity transient signals (HITS) representing solid or gaseous microembolism reaching the cerebral vessels.

Methods

Patients undergoing SAVR are included in the study and randomised to either MECC or CECC technique. HITS are continuously bilaterally detected during the entire intraoperative period by transcranial Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Severe Aortic Valve Stenosis
* No other cardiac disease
* No other coronary heart disease
* Written informed consent

Exclusion Criteria

* Double valve surgery
* Concomitant coronary artery bypass surgery
* Vascular surgery
* Age < 18 yrs.
* Age > 80 yrs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Total and interval-related cerebral microembolic load as measured by transcranial Doppler | Intraoperative period (start surgical procedure to skin suture, duration approx. 4 hrs)

SECONDARY OUTCOMES:
Cerebral complications, e.g. delirium and stroke as detected clinically | In-hospital period (until hospital discharge, duration approx. 7-10 days)
Redo surgery | In-hospital period (until hospital discharge, duration approx. 7-10 days)
ICU length of stay | In-hospital period (until hospital discharge, duration approx. 7-10 days)
Extubation time | In-hospital period (until hospital discharge, duration approx. 7-10 days)
Thromboembolic complications | In-hospital period (until hospital discharge, duration approx. 7-10 days)
In-hospital infections | In-hospital period (until hospital discharge, duration approx. 7-10 days)
In-hospital Mortality | In-hospital period (until hospital discharge, duration approx. 7-10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Carrel, MD, PhD, Principal Investigator — Department of Cardiovascular Surgery
Locations (1):
- University Hospital Bern, Bern, Switzerland